CLINICAL TRIAL: NCT04165681
Title: Evaluating the Feasibility of Limbix Spark: a Cognitive Behavioral Therapy Based Mobile and Virtual Reality Intervention for Adolescent Depression
Brief Title: A Mobile and Virtual Reality Intervention for Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Limbix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Limbix Spark 01
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Depression
Keywords: Adolescence; Cognitive Behavioral Therapy; Virtual Reality; Depression; Behavioral Activation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limbix Spark (Experimental): A 5 week mobile + virtual reality CBT-based program
  Interventions: Other: Limbix Spark

INTERVENTIONS:
Other: Limbix Spark — 5-week, self-guided mobile + VR CBT-based program for adolescent depression

SUMMARY:
Depression, the most common mental health disorder among adolescents, is a critical health problem within the US. In this study, the feasibility, acceptability, and preliminary efficacy of Limbix Spark, a cognitive behavioral therapy (CBT)- based mobile app + virtual reality (VR) program for helping adolescents live well with depression will be investigated. This program is specifically designed around behavioral activation theory, the idea that completing activities that make a patient feel pleasure or provide a sense of mastery are effective in reducing symptoms of depression. The program involves the use of both VR and a mobile app that include CBT components like psychological assessments, psychoeducation, and skills training. 30 participants aged 12-21 years old with mild to severe depressive symptoms and smartphone access will be enrolled in this study. The primary efficacy outcome measures will be depressive symptoms with anxiety symptoms, functional outcomes, and dimensional scales of positive and negative affect and behavioral activation serving as secondary outcome measures. Qualitative and quantitative feedback on the use of the VR + mobile app (ease of use, comfort, willingness to use again) will be assessed using questionnaires. Engagement and adherence to the program will be assessed by assessing VR and app usage.

DETAILED DESCRIPTION:
Depression, the most common mental health disorder among adolescents, is a major public health concern with significant personal, societal, and economic burdens, particularly as incidence rates are increasing. Effective care for adolescent depression is limited due to lack of access to care, increasingly long waitlists, stigma surrounding mental health, and ineffectiveness of pharmaceutical options. There is an urgent need for accessible, cost-effective, and evidence-based treatment options for adolescents with depression.

The development of effective digital health programs for adolescents is a key strategy to reduce the personal, familiar and societal burden of depression. Such programs provide an innovative way to deliver resources in a cost-effective, accessible fashion. Cognitive-behavioral therapy (CBT) is effective in the prevention and treatment of depression in children and adolescents. Digital forms of CBT have also been shown to be efficacious in the treatment of anxiety and depressive symptoms in youth, however. adherence to such programs in clinical trials and particularly in real world evidence evaluations is low. Virtual reality (VR) holds promise as a way to enhance adherence to and the efficacy of digital CBT for depression.

To address the need for effective, accessible, and engaging treatments for adolescent depression, the objective of this project is to evaluate the feasibility, acceptability, and preliminary evidence of efficacy of Limbix Spark: a 5 week CBT-based mobile + VR self-guided program. Limbix Spark is specifically designed to implement behavioral activation, a CBT skill, which involves completing self-monitored activities that provide a sense of pleasure or mastery in order to reduce depressive symptoms and improve functional outcomes. VR allows adolescents to complete such activities in virtual environments as a potential stepping stone to engaging in similar experiences in the real world.

30 participants aged 12-21 years old with mild to severe depressive symptoms and with smart phone access will be enrolled. During a baseline visit, participants or participants' legal guardians, will be asked to provide written informed consent and potential participants under 18 will be asked to provide written assent after study procedures are explained and any questions are answered by study staff in accordance with good clinical practice (GCP) and human subjects research guidelines.

After consent, all eligible participants will be assigned to complete the 5-week Limbix Spark program. Participants and their legal guardian if under 18 will first complete baseline assessments, including the Patient Health Questionnaire (PHQ-8) Generalized Anxiety Disorder scale (GAD-7), the Positive and Negative Affective Schedule (PANAS-C), the Behavioral Activation for Depression Scale-Short Form (BADS-SF), 20-item Short Form Survey (SF-20), Mood and Feelings Questionnaire Short Parent version (MFQ-PS). Participants will then receive VR equipment, and receive an initial orientation to the Limbix Spark program. Program orientation will include training on how to set up and use the VR headset and how to download and use the mobile app.

The 5 modules in the Limbix Spark program are meant to be completed weekly, however, participants will be allowed to progress through the program at their own pace. Each module contains VR and mobile app components and is expected to take no more than 60 minutes to complete, with no more than approximately 25 min per module of VR content. Modules do not need to be completed in a single session and can be completed over the course of several days. During the program, weekly PHQ-8 assessments will be completed within the mobile app.

At the post-intervention site visit, participants and their legal guardian if under 18 will complete post-program assessments, including the PHQ-8, GAD-7, PANAS-C, MFQ-PS, SF-20, and BADS-SF, as well as a questionnaire about their thoughts and experiences with the Spark program. Participants will also complete a qualitative interview to further understand their experience with the program.

One month after the post-intervention site visit, participants will be sent a 1-month follow up questionnaires via email, including the PHQ-8, GAD-7, PANAS-C, MFQ-PS, SF-20, and BADS-SF, as well as a questionnaire about their thoughts and experiences with the Spark program.

ELIGIBILITY:
Inclusion Criteria:

1. Score of 10 or greater on Patient Health Questionnaire (PHQ-8)
2. English fluency and literacy
3. Access to a smart phone
4. Patient willing to provide informed consent/assent and have parent/guardian willing to provide informed consent if under 18.

Exclusion Criteria:

1. Seizure disorder or other neurological disorder
2. Prior diagnosis of or receiving treatment for substance use disorder, bipolar disorder, or psychosis
3. Significant vision or hearing impairment
4. Hospitalized or received residential/inpatient treatment for a suicide attempt or self-harming behaviors within the past 3 months
5. Current diagnosis of a reading/learning or intellectual disability.
6. Receiving treatment (including but not limited to medication or psychotherapy) for a cognitive disorder, including attention deficit hyperactivity disorder (ADHD).
7. Are currently participating in a treatment study.
8. Pregnancy
9. History of significant motion sickness

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Adherence to program | Post treatment (5 weeks)
  % of enrolled participants completing all sessions at post treatment
Change in depression post treatment | Change from Baseline to Post treatment (5 weeks)
  Change in depressive symptoms measured by Personal Health Questionnaire (PHQ-8) (min: 0; max: 24, with higher score indicating more severe depression).

SECONDARY OUTCOMES:
Change in depression at one month follow up | Change from Baseline to 1 month follow up (9 weeks)
  Change in depressive symptoms measured by Personal Health Questionnaire (PHQ-8) (min: 0; max: 24, with higher score indicating more severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lake, PhD, Principal Investigator — Director of Research
Locations (1):
- Limbix Health, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller I, Peake E, Strauss G, Vierra E, Koepsell X, Shalchi B, Padmanabhan A, Lake J. Self-Guided Digital Intervention for Depression in Adolescents: Feasibility and Preliminary Efficacy Study. JMIR Form Res. 2023 Nov 22;7:e43260. doi: 10.2196/43260. PMID 37991839